CLINICAL TRIAL: NCT07227493
Title: Acute Bone Grafting of Open Pilon Fractures With FIBERGRAFT AERIDYAN Matrix Bioactive Glass
Brief Title: Open Pilon With FIBERGRAFT AERIDYAN Matrix Bioactive Glass
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Kyle Schweser MD, ASSOCIATE PROFESSOR OF ORTHOPAEDIC SURGERY, University of Missouri-Columbia
Other Study IDs: 2122307; 0081670 (Other Grant/Funding Number: DePuy Orthopaedics, Inc.)
Record Dates: First submitted 2025-06-18; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Open Pilon Fractures
Keywords: pilon; bone graft; open pilon; fibergraft; fibergraft aeridyan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Fibergraft Aeridyan Bone Graft Matrix: Patients in this group will be those who present to our institution with an open pilon fracture who receive the Fibergraft Aeridyan Bone Graft Matrix as part of their treatment for their pilon fracture.
  Interventions: Device: Fibergraft Aeridyan Matrix

INTERVENTIONS:
Device: Fibergraft Aeridyan Matrix — FIBERGRAFT™ Aeridyan™ Matrix is a resorbable porous bone graft substitute made from 45S5 bioactive glass, boron bioactive glass and type I collagen. The implantable material is provided as a premixed Matrix of bioactive granules and microspheres in a collagen carrier.

SUMMARY:
Open pilon fractures are challenging problems to manage. Infection rates vary from 6-30% and metaphyseal nonunion varies from 7-20%. The current recommendation for the management of open pilon fractures with bone loss is a staged approach, with internal fixation around an antibiotic spacer. Fibergraft Aeridyan Bone Graft Matrix is currently used along with other forms of allograft at our institution for filling bone voids in open pilon fractures. This is a prospective, observational study looking at the use of Fibergraft Aeridyan bone graft matrix and its efficacy in open pilon fractures. Everything in this study will be according to the standard of care at our institution other than two research only CT scans. One will be performed at the patient's 6-month visit and the other will be performed at the patient's 12-month visit. The investigators hypothesize that Fibergraft Aeridyan Bone Graft Matrix will lead to improved outcomes when compared to standard bone graft for patients by decreasing infection and nonunion rates.

DETAILED DESCRIPTION:
Tibial plafond, or pilon fractures are complicated, rare, challenging fractures representing less than 1% of all lower extremity fractures and 1-10% of all tibial fractures.1 A quarter of these pilon fractures are open and involve soft tissue complications and could lead to amputation if not treated properly.1-3

The AO/OTA classifies these pilon fractures as 43A-C,1-34; and are often open fractures characterized by the Gustilo Anderson (GA) scale.5 These high energy traumatic injuries are often susceptible to multiple complications such as superficial infection, fracture related infection, and non-union.1,2,6,7

There are a variety of surgical incisional approaches that depend on the type and kind of pilon fracture and are often a staged procedure relative to the soft tissue trauma, edema, vascularization, and the surgeon's experience.1,8,9 Open pilon fractures are challenging problems to manage. Infection rates vary from 6-30% and metaphyseal nonunion varies from 7-20%.

The current recommendation for the management of open pilon fractures with bone loss is a staged approach, with internal fixation around an antibiotic spacer. Some studies have examined the use of acute allograft with BMP for larger defects, however, the success rate was variable. Several issues exist when it comes to acute bone grafting of open pilon fractures. The first is that the bone defect is often too large for autograft secondary to comminution of the remaining tibia, and metaphyseal impaction, around the area of bone loss. This requires more bone graft than returning later once secondary bone healing has begun to occur. The second is the concern for deep infections, which is relatively high when compared to other open fractures. Introducing allograft bone is concerning for patients who are already at a high risk of infection. The third is soft tissue concerns. The open laceration is most commonly on the anteromedial/medial side of the tibia and occurs via tension on the skin. This sheering force on the tissue causes significant disruption of the surrounding microvasculature, causing delayed wound healing, limited delivery of antibiotics, and potentially contributes to the higher rate of nonunion in the tibial metaphysis. Aeridyan has the potential to overcome several of these concerns secondary to its ability to fill a larger void, improve the microenvironment for healing by osteoblast proliferation, improve blood flow through its angiogenic properties, and decrease risk of infection secondary to its potential bactericidal properties. These benefits, among others, may improve rates of healing (decreasing the nonunion rates) and decrease secondary surgeries (return for planned bone grafting/deep infections).

The primary objective will be the radiographic healing (mRUST average grade 6-8) of open pilon fractures after application of FIBERGRAFT AERIDYAN Matrix bioactive glass and ORIF at 12 months. The secondary objectives will be looking at wound healing complications, infection rates, and unplanned secondary operations and radiographic healing of open pilon fractures after application of FIBERGRAFT AERIDYAN Matrix bioactive glass and ORIF at 6 months.

Current complication rates associated with pilon fractures using bone graft include a high metaphyseal nonunion rate (7-20%) and a high infection rate (6-30%). The Investigators hypothesize that Fibergraft Aeridyan Bone Graft Matrix will lead to improved outcomes when compared to standard bone graft for patients by decreasing infection and nonunion rates. The use of Aeridyan will be compared to the already well-reported outcomes in the literature regarding the use of bone grafting with open reduction and internal fixation (ORIF) for pilon fractures. All adverse events will be tracked and reported to DePuy Orthopaedics as complaints. Should there be a serious adverse event that is device related, then the subject will discontinue the study.

The FDA classifies Fibergraft Aeridyan Bone Graft Matrix as a class II medical device, and the FDA has provided 510(K) clearance for this device.

Patients will be screened in either the orthopaedic trauma clinic or preoperatively for patients who present to the hospital with a trauma and an open pilon fracture who require fixation with ORIF and bone grafting. If determined to meet all inclusion criteria, the patient will be approached by the surgeon or a member of the research team to obtain voluntary informed consent.

A member of the research team will consent the study candidate prior to definitive care while they are in-patient or prior to surgery while they at the University of Missouri Hospital/Missouri Orthopaedic Institute. The research study, protocol, and consent will be thoroughly explained, and all questions will be answered in a private setting. Once all questions have been answered and the candidate demonstrates full understanding, the candidate will be asked to sign the consent form with HIPPA Authorization. They will be given a copy of the consent form to keep with them and are able to ask questions as they arise.

The Investigators anticipate enrolling 45 participants over a 3-year time period. Pilon fractures are complicated, rare, challenging fractures representing less than 1% of all lower extremity fractures. Numbers were selected based on feasibility of study completion for a prospective cohort study in 3 years over 1 site. This number of subjects will allow for adequate data collection and comparison to the current literature regarding treatment of open pilon fractures.

This is a prospective cohort study of open pilon fractures. Patients presenting with open pilon fractures will receive the standard of care for the institution in terms of antibiotics, tetanus, wound care, and splinting. Patients will then undergo external fixation. During the initial surgery, if any bone is removed, this will be quantified and documented. During the initial external fixation, antibiotic beads or cement may be utilized as a void filler while awaiting definitive surgery. If bone loss requiring bone grafting is noted on the initial x-rays, initial surgical findings, or post operative CT scan, then patients will be screened and enrolled in the study upon providing consent. Patients requiring multiple irrigation and debridement procedures and those requiring flap coverage will remain enrolled in the study. Patients will undergo the standard of care for management of open pilon fractures up until definitive fixation. Definitive fixation will occur at the discretion of the managing surgeon, typically occurring within 10-14 days from application of the external fixator. A post operative CT scan will be utilized to calculate the area of bone loss, and at 6 months and then 12 months. At the time of definitive fixation, the bone void will be measured to allow for a secondary calculation of bone loss, and Aeridyan matrix, which is currently already being used as standard of care, will be utilized to fill the void. The amount will be recorded. Patients will then be closed at the discretion of the managing physician. Post-operatively, patients will be seen in clinic at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months. Any wound complication and action taken will be recorded. X-rays will be taken at 6 weeks, 3 months, 6 months, and 12 months. Patient reported outcomes (PROMIS PF, AAOS foot and ankle) will be collected at each post operative visit. Weightbearing will be up to the discretion of the treating surgeon. A CT scan will be obtained at 6 and 12 months to assess healing of the bone void. Any return trip to the operating room will be documented.

Research only (non-standard of care) interventions:

• Post-operative CT scans at the standard of care 6- and 12-month visits to calculate the area of bone loss

There will be no blinding in this study. All enrolled participants will receive the Aeridyan matrix. Results will be compared to the well documented results in the literature regarding the use of bone grafting during ORIF of open pilon fractures.

There is minimal risk with breach of confidential medical information. Efforts will be made to avoid the breach of confidentiality. Records are given a study identification number that will be free of subject's name and identifiers. Identification numbers connected with subjects' names will be kept in a secure location and otherwise will be archived in a secure storage facility or destroyed. All risks would be similar or equal to standard of care as they involve implantation of rigid fixation, and the inherent risks of surgery. Adverse events to be collected will be associated with device and open pilon fractures: fracture nonunion, fracture related infection, pin tract infection, soft tissue infection, unexpected wound exudate or fluid buildup, hardware failure and re-operation and will be observed/treated by the investigator as part of the standard of care treatment. CT scans expose patients to radiation similar to x-rays. Additionally, CT scans may make patients feel uncomfortable while undergoing testing.

Subject safety will be ensured through standard of care procedures and monitoring by clinical and surgical staff. Data will be recorded on paper source documents for the various endpoints, with data verification occurring a time of entry into EDC. PROs are directly entered into Patient IQ by the participant. Patient IQ contains INPUT validations to ensure data integrity. A sequential 1-30 patient number will be assigned instead of personally identifiable information. There will be a subject enrollment log with corresponding MRN/ID number-key that only the investigator and study staff will retain to link the patient records to the study case report forms. Paper source documents will be stored in a locked cabinet/room with only approved staff having access. Electronic medical records (CERNER) will be the primary source document with all associated security; data transposed into Patient IQ using defined case report forms for clinical study. Patient IQ is a cloud-based HIPAA Compliant, HITRUST CSF Certified, 21 CFT Part 11 Compliant platform used to collect patient reported outcomes and data containing built in INPUT validations to ensure data integrity.

The Principal Investigator (PI) will monitor the study for safety, with a focus on serious adverse events (SAEs) and unexpected reactions related to the Fibergraft Aeridyan Matrix Bioactive Glass product. These events will be monitored as part of standard of care treatment as they occur.

The PI will adapt monitoring based on emerging risks and ensure ongoing communication with the study team and sponsor, providing regular reports and addressing any urgent safety issues. All actions and decisions will be documented and shared with the sponsor to ensure patient safety and trial integrity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Open pilon fracture requiring bone grafting
* Able to provide informed consent for the study prior to definitive care

Exclusion Criteria:

* Under 18 years of age
* Open pilon fracture not requiring bone grafting
* Receiving definitive care at an outside facility
* Unlikely to make follow-up appointments
* Active infection at the time of definitive care
* Unable to provide informed consent prior to definitive care
* Prisoners
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to our institution with an open pilon fracture that will undergo open reduction with internal fixation and will require bone grafting.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The number of participants that demonstrate radiographic healing at 12 months, as assessed by the mRUST | 12 months
  Participants will be assessed for radiographic healing through a modified radiographic union score for tibial fractures (mRUST), with an average grade of 6-8 per radiograph after application of FIBERGRAFT AERIDYAN Matrix bioactive glass and ORIF at 12 months.
  mRUST is scored on a scale of 1-4 for each cortex. 1: no callus is present, 2: callus is present, 3: bridging callus is present, 4: fracture line is no longer visible. 2 cortices are visible per radiographic image. Therefore, there is a max score of 8 per radiograph. Scores with an average of 6-8 in this study are deemed as demonstrating radiographic healing.

SECONDARY OUTCOMES:
The number of participants that experience wound complications, as assessed by a part of standard of care treatment | 12 months
  Participants will be assessed for wound complications, such as delayed wound healing, wound dehiscence, infection, and unplanned secondary operations, through standard of care wound checks at follow-up visits.
The number of participants that demonstrate radiographic healing at 6 months, as assessed by the mRUST | 6 months
  Participants will be assessed for radiographic healing through a modified radiographic union score for tibial fractures (mRUST), with an average grade of 6-8 per radiograph after application of FIBERGRAFT AERIDYAN Matrix bioactive glass and ORIF at 6 months.
  mRUST is scored on a scale of 1-4 for each cortex. 1: no callus is present, 2: callus is present, 3: bridging callus is present, 4: fracture line is no longer visible. 2 cortices are visible per radiographic image. Therefore, there is a max score of 8 per radiograph. Scores with an average of 6-8 in this study are deemed as demonstrating radiographic healing.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Schweser, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

REFERENCES:
- [Background] Ziegenhain F, Neuhaus V, Pape HC. Bioactive glass in the treatment of chronic osteomyelitis-a valid option? OTA Int. 2021 Jun 15;4(3 Suppl):e105(1-4). doi: 10.1097/OI9.0000000000000105. eCollection 2021 Jun. PMID 37609479
- [Background] Waltimo T, Brunner TJ, Vollenweider M, Stark WJ, Zehnder M. Antimicrobial effect of nanometric bioactive glass 45S5. J Dent Res. 2007 Aug;86(8):754-7. doi: 10.1177/154405910708600813. PMID 17652205
- [Background] Fiume E, Barberi J, Verne E, Baino F. Bioactive Glasses: From Parent 45S5 Composition to Scaffold-Assisted Tissue-Healing Therapies. J Funct Biomater. 2018 Mar 16;9(1):24. doi: 10.3390/jfb9010024. PMID 29547544
- [Background] Zimmermann G, Moghaddam A. Allograft bone matrix versus synthetic bone graft substitutes. Injury. 2011 Sep;42 Suppl 2:S16-21. doi: 10.1016/j.injury.2011.06.199. Epub 2011 Sep 1. PMID 21889142
- [Background] Kim WY, Ji JH, Park SE, Kim YY, Jeong JJ, Kang HT. Surgical management of pilon fractures with large segmental bone defects using fibular strut allografts: a report of two cases. Eur J Orthop Surg Traumatol. 2011 Aug;21(6):439-444. doi: 10.1007/s00590-010-0732-3. Epub 2011 Mar 25. PMID 21874131
- [Background] Meng YC, Zhou XH. External fixation versus open reduction and internal fixation for tibial pilon fractures: A meta-analysis based on observational studies. Chin J Traumatol. 2016 Oct 1;19(5):278-282. doi: 10.1016/j.cjtee.2016.06.002. PMID 27780508
- [Background] Carter TH, Duckworth AD, Oliver WM, Molyneux SG, Amin AK, White TO. Open Reduction and Internal Fixation of Distal Tibial Pilon Fractures. JBJS Essent Surg Tech. 2019 Sep 11;9(3):e29. doi: 10.2106/JBJS.ST.18.00093. eCollection 2019 Jul-Sep. PMID 32021729
- [Background] Korkmaz A, Ciftdemir M, Ozcan M, Copuroglu C, Saridogan K. The analysis of the variables, affecting outcome in surgically treated tibia pilon fractured patients. Injury. 2013 Oct;44(10):1270-4. doi: 10.1016/j.injury.2013.06.016. Epub 2013 Jul 18. PMID 23871428
- [Background] Gustilo RB, Gruninger RP, Davis T. Classification of type III (severe) open fractures relative to treatment and results. Orthopedics. 1987 Dec;10(12):1781-8. PMID 3324085
- [Background] Bear J, Rollick N, Helfet D. Evolution in Management of Tibial Pilon Fractures. Curr Rev Musculoskelet Med. 2018 Dec;11(4):537-545. doi: 10.1007/s12178-018-9519-7. PMID 30343399
- [Background] Mauffrey C, Vasario G, Battiston B, Lewis C, Beazley J, Seligson D. Tibial pilon fractures: a review of incidence, diagnosis, treatment, and complications. Acta Orthop Belg. 2011 Aug;77(4):432-40. PMID 21954749
- [Background] Kugach KA, Leong WM, Clements JR. Management of Pilon Fractures. Clin Podiatr Med Surg. 2024 Jul;41(3):503-518. doi: 10.1016/j.cpm.2024.01.007. Epub 2024 Feb 28. PMID 38789167